CLINICAL TRIAL: NCT05989126
Title: A Study in Patients With Diabetic Macular Edema or Neovascular Age-Related Macular Degeneration to Evaluate a High Dose Aflibercept (8 mg) Prefilled Syringe
Brief Title: Study to Evaluate an 8 mg Aflibercept (EYLEA®) Prefilled Syringe (PFS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-HD-OD-22105
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Macular Edema (DME); Neovascular Age-Related Macular Degeneration (nAMD)
Keywords: Neovascular "wet" age-related macular degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 8 mg Dose (Experimental): Only 1 eye will be selected as the study eye by the investigator. Patients will receive a single dose utilizing the PFS.
  Interventions: Drug: aflibercept 8 mg PFS

INTERVENTIONS:
Drug: aflibercept 8 mg PFS — Sterile aqueous solution in a single-dose PFS administered by intravitreal (IVT) injection
  Other Names: EYLEA ® HD; BAY86-5321

SUMMARY:
Regeneron Pharmaceuticals developed a single-dose pre-filled syringe (PFS) to deliver 8 mg aflibercept. The PFS is a convenient device that contains the study medication that will be injected in your study eye. A PFS offers a sterile, single dose of study drug within the syringe; this eliminates the need for the retina specialist to prepare the injection syringe from a separate vial.

This Phase IIIb study is focused on patients with diabetic macular edema (DME) and neovascular (wet) age-related macular degeneration (nAMD).

The main aim of the study is to evaluate if the 8 mg aflibercept PFS allows for successful preparation and administration of 8 mg aflibercept by retina specialists. The study will also assess the safety of 8 mg aflibercept PFS use. Regeneron will use the information from the study to better understand if the PFS can be used safely and effectively by retina specialists to administer 8 mg aflibercept.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patient must have diabetic macular edema (DME) or neovascular "wet" age-related macular degeneration (nAMD) in the study eye
2. Study eye considered by the retina specialist to be eligible for treatment with 8 mg aflibercept

Key Exclusion Criteria:

1. Any active intraocular inflammation or infection in either eye or history of intraocular inflammation or infection after past IVT injections with any agent in either eye
2. Treatment with any IVT injection in the study eye within the 25 days prior to day 1
3. Intraocular pressure (IOP) >25 mm Hg in the study eye at screening
4. Any intraocular surgery in the study eye at any time during the past 3 months
5. Any prior extended-release therapeutic agent, or ocular drug-release device implantation (approved or investigational, including steroids) in the study eye

NOTE: Other protocol Defined Inclusion/Exclusion Criteria Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Number of 8 mg aflibercept injections successfully administered utilizing the PFS | At Day 1
  Participants received a single dose of study drug, administered in the selected study eye with the PFS by a retina specialist. Physician assessed successful aflibercept preparation and administration with the PFS.

SECONDARY OUTCOMES:
Incidence of ocular adverse events (AEs) in the study eye | Through Day 29
Incidence of ocular severe adverse events (SAEs) in the study eye | Through Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/